CLINICAL TRIAL: NCT04872036
Title: Investigation of Prognostic Biomarkers in Patients With Urothelial Carcinoma Treated With Platinum Regimens
Brief Title: Prognostic Biomarkers in Patients With Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: Biomarkers_Urothelial
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Bladder Cancer
Keywords: Next Generation sequencing; TP53; ARID1A; ERCC2; BRACA2; DNA damage response; platinum sensitivity; muscle invasive; PD-L1; CD8; TILs; MMR
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder cancer (BC) is a heterogeneous malignancy with dismal outcome.Despite treatment, the 5-year overall survival rates for MIBC are <50%, with many patients unresponsive or inapt, necessitating biomarkers to select those most likely to respond or fit for treatment

DETAILED DESCRIPTION:
In this study was assessed the associations among most frequently mutated genes and with clinicopathological features, as well as the prognostic significance of the presence of mutations in the top mutated and DNA Damage response (DDR) mutated genes in terms of Overall Survival (OS). Moreover, overall tumor-infiltrating lymphocytes (TILs) density was measured, analyzed immunohistochemically the expression of PD-L1, the four MMR proteins (MLH1, MSH2, MSH6 and PMS2) and tumor or stromal CD8+ cytotoxic T lymphocyte infiltrates and assessed their association with each other, top mutated genes and available clinicopathological parameters together with their role in prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Urothelial carcinoma located in bladder
* Patients treated with platinum regimens at the neoadjuvant . adjuvant setting
* Written informed consent for the use of biological material

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a transnational analysis with biosamples from patients with urothelial carcinoma treated with platinum regimes. Patients have been treated in Hellenic Cooperative Oncology Group (HeCOG) affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of mutational profile in patients with urothelial carcinoma | Up to 5 years

SECONDARY OUTCOMES:
Association of mutational profile with PD-L1 expression | Up to 5 years
Association of the prognostic significance of mutations with respect to overall survival | Up to 5 years

REFERENCES:
- [Background] Soria F, Krabbe LM, Todenhofer T, Dobruch J, Mitra AP, Inman BA, Gust KM, Lotan Y, Shariat SF. Molecular markers in bladder cancer. World J Urol. 2019 Jan;37(1):31-40. doi: 10.1007/s00345-018-2503-4. Epub 2018 Sep 26. PMID 30259123
- [Background] https://www.intechopen.com/books/bladder-cancer-management-of-nmi-and-muscle-invasive-cancer/bladder-cancer-markers-and-recent-innovations
- [Background] Solomon JP, Hansel DE. The Emerging Molecular Landscape of Urothelial Carcinoma. Surg Pathol Clin. 2016 Sep;9(3):391-404. doi: 10.1016/j.path.2016.04.004. PMID 27523968
- [Background] Koga F, Takemura K, Fukushima H. Biomarkers for Predicting Clinical Outcomes of Chemoradiation-Based Bladder Preservation Therapy for Muscle-Invasive Bladder Cancer. Int J Mol Sci. 2018 Sep 15;19(9):2777. doi: 10.3390/ijms19092777. PMID 30223570
- [Background] Apollo A, Ortenzi V, Scatena C, Zavaglia K, Aretini P, Lessi F, Franceschi S, Tomei S, Sepich CA, Viacava P, Mazzanti CM, Naccarato AG. Molecular characterization of low grade and high grade bladder cancer. PLoS One. 2019 Jan 16;14(1):e0210635. doi: 10.1371/journal.pone.0210635. eCollection 2019. PMID 30650148
- [Background] Guo CC, Czerniak B. Bladder Cancer in the Genomic Era. Arch Pathol Lab Med. 2019 Jun;143(6):695-704. doi: 10.5858/arpa.2018-0329-RA. Epub 2019 Jan 23. PMID 30672335
- [Background] Chandrasekar T, Erlich A, Zlotta AR. Molecular Characterization of Bladder Cancer. Curr Urol Rep. 2018 Nov 3;19(12):107. doi: 10.1007/s11934-018-0853-5. PMID 30390141
- [Background] Matulay JT, Kamat AM. Advances in risk stratification of bladder cancer to guide personalized medicine. F1000Res. 2018 Jul 25;7:F1000 Faculty Rev-1137. doi: 10.12688/f1000research.14903.1. eCollection 2018. PMID 30109022
- [Background] Song YP, McWilliam A, Hoskin PJ, Choudhury A. Organ preservation in bladder cancer: an opportunity for truly personalized treatment. Nat Rev Urol. 2019 Sep;16(9):511-522. doi: 10.1038/s41585-019-0199-x. Epub 2019 Jun 13. PMID 31197260
- [Background] Pardo JC, Ruiz de Porras V, Plaja A, Carrato C, Etxaniz O, Buisan O, Font A. Moving towards Personalized Medicine in Muscle-Invasive Bladder Cancer: Where Are We Now and Where Are We Going? Int J Mol Sci. 2020 Aug 29;21(17):6271. doi: 10.3390/ijms21176271. PMID 32872531
- [Background] Choi W, Porten S, Kim S, Willis D, Plimack ER, Hoffman-Censits J, Roth B, Cheng T, Tran M, Lee IL, Melquist J, Bondaruk J, Majewski T, Zhang S, Pretzsch S, Baggerly K, Siefker-Radtke A, Czerniak B, Dinney CP, McConkey DJ. Identification of distinct basal and luminal subtypes of muscle-invasive bladder cancer with different sensitivities to frontline chemotherapy. Cancer Cell. 2014 Feb 10;25(2):152-65. doi: 10.1016/j.ccr.2014.01.009. PMID 24525232
- [Background] Robertson AG, Kim J, Al-Ahmadie H, Bellmunt J, Guo G, Cherniack AD, Hinoue T, Laird PW, Hoadley KA, Akbani R, Castro MAA, Gibb EA, Kanchi RS, Gordenin DA, Shukla SA, Sanchez-Vega F, Hansel DE, Czerniak BA, Reuter VE, Su X, de Sa Carvalho B, Chagas VS, Mungall KL, Sadeghi S, Pedamallu CS, Lu Y, Klimczak LJ, Zhang J, Choo C, Ojesina AI, Bullman S, Leraas KM, Lichtenberg TM, Wu CJ, Schultz N, Getz G, Meyerson M, Mills GB, McConkey DJ; TCGA Research Network; Weinstein JN, Kwiatkowski DJ, Lerner SP. Comprehensive Molecular Characterization of Muscle-Invasive Bladder Cancer. Cell. 2017 Oct 19;171(3):540-556.e25. doi: 10.1016/j.cell.2017.09.007. Epub 2017 Oct 5. PMID 28988769
- [Background] Choi W, Ochoa A, McConkey DJ, Aine M, Hoglund M, Kim WY, Real FX, Kiltie AE, Milsom I, Dyrskjot L, Lerner SP. Genetic Alterations in the Molecular Subtypes of Bladder Cancer: Illustration in the Cancer Genome Atlas Dataset. Eur Urol. 2017 Sep;72(3):354-365. doi: 10.1016/j.eururo.2017.03.010. Epub 2017 Mar 30. PMID 28365159
- [Background] Guo G, Sun X, Chen C, Wu S, Huang P, Li Z, Dean M, Huang Y, Jia W, Zhou Q, Tang A, Yang Z, Li X, Song P, Zhao X, Ye R, Zhang S, Lin Z, Qi M, Wan S, Xie L, Fan F, Nickerson ML, Zou X, Hu X, Xing L, Lv Z, Mei H, Gao S, Liang C, Gao Z, Lu J, Yu Y, Liu C, Li L, Fang X, Jiang Z, Yang J, Li C, Zhao X, Chen J, Zhang F, Lai Y, Lin Z, Zhou F, Chen H, Chan HC, Tsang S, Theodorescu D, Li Y, Zhang X, Wang J, Yang H, Gui Y, Wang J, Cai Z. Whole-genome and whole-exome sequencing of bladder cancer identifies frequent alterations in genes involved in sister chromatid cohesion and segregation. Nat Genet. 2013 Dec;45(12):1459-63. doi: 10.1038/ng.2798. Epub 2013 Oct 13. PMID 24121792
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of urothelial bladder carcinoma. Nature. 2014 Mar 20;507(7492):315-22. doi: 10.1038/nature12965. Epub 2014 Jan 29. PMID 24476821
- [Background] Audenet F, Attalla K, Sfakianos JP. The evolution of bladder cancer genomics: What have we learned and how can we use it? Urol Oncol. 2018 Jul;36(7):313-320. doi: 10.1016/j.urolonc.2018.02.017. Epub 2018 Mar 21. PMID 29573965
- [Background] Heeke AL, Pishvaian MJ, Lynce F, Xiu J, Brody JR, Chen WJ, Baker TM, Marshall JL, Isaacs C. Prevalence of Homologous Recombination-Related Gene Mutations Across Multiple Cancer Types. JCO Precis Oncol. 2018;2018:PO.17.00286. doi: 10.1200/PO.17.00286. Epub 2018 Jul 23. PMID 30234181
- [Background] Abbosh PH, Plimack ER. Molecular and Clinical Insights into the Role and Significance of Mutated DNA Repair Genes in Bladder Cancer. Bladder Cancer. 2018 Jan 20;4(1):9-18. doi: 10.3233/BLC-170129. PMID 29430503
- [Background] Yap KL, Kiyotani K, Tamura K, Antic T, Jang M, Montoya M, Campanile A, Yew PY, Ganshert C, Fujioka T, Steinberg GD, O'Donnell PH, Nakamura Y. Whole-exome sequencing of muscle-invasive bladder cancer identifies recurrent mutations of UNC5C and prognostic importance of DNA repair gene mutations on survival. Clin Cancer Res. 2014 Dec 15;20(24):6605-17. doi: 10.1158/1078-0432.CCR-14-0257. Epub 2014 Oct 14. PMID 25316812
- [Background] Liu D, Plimack ER, Hoffman-Censits J, Garraway LA, Bellmunt J, Van Allen E, Rosenberg JE. Clinical Validation of Chemotherapy Response Biomarker ERCC2 in Muscle-Invasive Urothelial Bladder Carcinoma. JAMA Oncol. 2016 Aug 1;2(8):1094-6. doi: 10.1001/jamaoncol.2016.1056. No abstract available. PMID 27310333
- [Background] Teo MY, Bambury RM, Zabor EC, Jordan E, Al-Ahmadie H, Boyd ME, Bouvier N, Mullane SA, Cha EK, Roper N, Ostrovnaya I, Hyman DM, Bochner BH, Arcila ME, Solit DB, Berger MF, Bajorin DF, Bellmunt J, Iyer G, Rosenberg JE. DNA Damage Response and Repair Gene Alterations Are Associated with Improved Survival in Patients with Platinum-Treated Advanced Urothelial Carcinoma. Clin Cancer Res. 2017 Jul 15;23(14):3610-3618. doi: 10.1158/1078-0432.CCR-16-2520. Epub 2017 Jan 30. PMID 28137924
- [Background] Teo MY, Seier K, Ostrovnaya I, Regazzi AM, Kania BE, Moran MM, Cipolla CK, Bluth MJ, Chaim J, Al-Ahmadie H, Snyder A, Carlo MI, Solit DB, Berger MF, Funt S, Wolchok JD, Iyer G, Bajorin DF, Callahan MK, Rosenberg JE. Alterations in DNA Damage Response and Repair Genes as Potential Marker of Clinical Benefit From PD-1/PD-L1 Blockade in Advanced Urothelial Cancers. J Clin Oncol. 2018 Jun 10;36(17):1685-1694. doi: 10.1200/JCO.2017.75.7740. Epub 2018 Feb 28. PMID 29489427
- [Background] Eckstein M, Cimadamore A, Hartmann A, Lopez-Beltran A, Cheng L, Scarpelli M, Montironi R, Gevaert T. PD-L1 assessment in urothelial carcinoma: a practical approach. Ann Transl Med. 2019 Nov;7(22):690. doi: 10.21037/atm.2019.10.24. PMID 31930091
- [Background] Hodgson A, Vesprini D, Liu SK, Xu B, Downes MR. Correlation of mismatch repair protein deficiency, PD-L1 and CD8 expression in high-grade urothelial carcinoma of the bladder. J Clin Pathol. 2020 Aug;73(8):519-522. doi: 10.1136/jclinpath-2019-206256. Epub 2020 Jan 9. PMID 31919144
- [Background] Wahlin S, Nodin B, Leandersson K, Boman K, Jirstrom K. Clinical impact of T cells, B cells and the PD-1/PD-L1 pathway in muscle invasive bladder cancer: a comparative study of transurethral resection and cystectomy specimens. Oncoimmunology. 2019 Aug 3;8(11):e1644108. doi: 10.1080/2162402X.2019.1644108. eCollection 2019. PMID 31646091
- [Background] Erlmeier F, Seitz AK, Hatzichristodoulou G, Stecher L, Retz M, Gschwend JE, Weichert W, Kubler HR, Horn T. The Role of PD-L1 Expression and Intratumoral Lymphocytes in Response to Perioperative Chemotherapy for Urothelial Carcinoma. Bladder Cancer. 2016 Oct 27;2(4):425-432. doi: 10.3233/BLC-160067. PMID 28035323
- [Background] Faraj SF, Munari E, Guner G, Taube J, Anders R, Hicks J, Meeker A, Schoenberg M, Bivalacqua T, Drake C, Netto GJ. Assessment of tumoral PD-L1 expression and intratumoral CD8+ T cells in urothelial carcinoma. Urology. 2015 Mar;85(3):703.e1-6. doi: 10.1016/j.urology.2014.10.020. PMID 25733301
- [Background] Balbas-Martinez C, Sagrera A, Carrillo-de-Santa-Pau E, Earl J, Marquez M, Vazquez M, Lapi E, Castro-Giner F, Beltran S, Bayes M, Carrato A, Cigudosa JC, Dominguez O, Gut M, Herranz J, Juanpere N, Kogevinas M, Langa X, Lopez-Knowles E, Lorente JA, Lloreta J, Pisano DG, Richart L, Rico D, Salgado RN, Tardon A, Chanock S, Heath S, Valencia A, Losada A, Gut I, Malats N, Real FX. Recurrent inactivation of STAG2 in bladder cancer is not associated with aneuploidy. Nat Genet. 2013 Dec;45(12):1464-9. doi: 10.1038/ng.2799. Epub 2013 Oct 13. PMID 24121791
- [Background] Kotoula V, Lakis S, Tikas I, Giannoulatou E, Lazaridis G, Papadopoulou K, Manoussou K, Efstratiou I, Papanikolaou A, Fostira F, Vlachos I, Tarlatzis B, Fountzilas G. Pathogenic BRCA1 mutations may be necessary but not sufficient for tissue genomic heterogeneity: Deep sequencing data from ovarian cancer patients. Gynecol Oncol. 2019 Feb;152(2):375-386. doi: 10.1016/j.ygyno.2018.11.016. Epub 2018 Nov 14. PMID 30446274
- [Background] Balar AV, Castellano D, O'Donnell PH, Grivas P, Vuky J, Powles T, Plimack ER, Hahn NM, de Wit R, Pang L, Savage MJ, Perini RF, Keefe SM, Bajorin D, Bellmunt J. First-line pembrolizumab in cisplatin-ineligible patients with locally advanced and unresectable or metastatic urothelial cancer (KEYNOTE-052): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Nov;18(11):1483-1492. doi: 10.1016/S1470-2045(17)30616-2. Epub 2017 Sep 26. PMID 28967485
- [Background] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060
- [Background] Bouaoun L, Sonkin D, Ardin M, Hollstein M, Byrnes G, Zavadil J, Olivier M. TP53 Variations in Human Cancers: New Lessons from the IARC TP53 Database and Genomics Data. Hum Mutat. 2016 Sep;37(9):865-76. doi: 10.1002/humu.23035. Epub 2016 Jul 8. PMID 27328919
- [Background] Chang MT, Asthana S, Gao SP, Lee BH, Chapman JS, Kandoth C, Gao J, Socci ND, Solit DB, Olshen AB, Schultz N, Taylor BS. Identifying recurrent mutations in cancer reveals widespread lineage diversity and mutational specificity. Nat Biotechnol. 2016 Feb;34(2):155-63. doi: 10.1038/nbt.3391. Epub 2015 Nov 30. PMID 26619011
- [Background] Chang MT, Bhattarai TS, Schram AM, Bielski CM, Donoghue MTA, Jonsson P, Chakravarty D, Phillips S, Kandoth C, Penson A, Gorelick A, Shamu T, Patel S, Harris C, Gao J, Sumer SO, Kundra R, Razavi P, Li BT, Reales DN, Socci ND, Jayakumaran G, Zehir A, Benayed R, Arcila ME, Chandarlapaty S, Ladanyi M, Schultz N, Baselga J, Berger MF, Rosen N, Solit DB, Hyman DM, Taylor BS. Accelerating Discovery of Functional Mutant Alleles in Cancer. Cancer Discov. 2018 Feb;8(2):174-183. doi: 10.1158/2159-8290.CD-17-0321. Epub 2017 Dec 15. PMID 29247016
- [Background] Baugh EH, Ke H, Levine AJ, Bonneau RA, Chan CS. Why are there hotspot mutations in the TP53 gene in human cancers? Cell Death Differ. 2018 Jan;25(1):154-160. doi: 10.1038/cdd.2017.180. Epub 2017 Nov 3. PMID 29099487
- [Background] Cleaver JE, Lam ET, Revet I. Disorders of nucleotide excision repair: the genetic and molecular basis of heterogeneity. Nat Rev Genet. 2009 Nov;10(11):756-68. doi: 10.1038/nrg2663. Epub 2009 Oct 7. PMID 19809470
- [Background] Van Allen EM, Mouw KW, Kim P, Iyer G, Wagle N, Al-Ahmadie H, Zhu C, Ostrovnaya I, Kryukov GV, O'Connor KW, Sfakianos J, Garcia-Grossman I, Kim J, Guancial EA, Bambury R, Bahl S, Gupta N, Farlow D, Qu A, Signoretti S, Barletta JA, Reuter V, Boehm J, Lawrence M, Getz G, Kantoff P, Bochner BH, Choueiri TK, Bajorin DF, Solit DB, Gabriel S, D'Andrea A, Garraway LA, Rosenberg JE. Somatic ERCC2 mutations correlate with cisplatin sensitivity in muscle-invasive urothelial carcinoma. Cancer Discov. 2014 Oct;4(10):1140-53. doi: 10.1158/2159-8290.CD-14-0623. Epub 2014 Aug 5. PMID 25096233
- [Background] Li Q, Damish AW, Frazier Z, Liu D, Reznichenko E, Kamburov A, Bell A, Zhao H, Jordan EJ, Gao SP, Ma J, Abbosh PH, Bellmunt J, Plimack ER, Lazaro JB, Solit DB, Bajorin D, Rosenberg JE, D'Andrea AD, Riaz N, Van Allen EM, Iyer G, Mouw KW. ERCC2 Helicase Domain Mutations Confer Nucleotide Excision Repair Deficiency and Drive Cisplatin Sensitivity in Muscle-Invasive Bladder Cancer. Clin Cancer Res. 2019 Feb 1;25(3):977-988. doi: 10.1158/1078-0432.CCR-18-1001. Epub 2018 Jul 6. PMID 29980530
- [Background] Mendiratta P, Grivas P. Emerging biomarkers and targeted therapies in urothelial carcinoma. Ann Transl Med. 2018 Jun;6(12):250. doi: 10.21037/atm.2018.05.49. PMID 30069452
- [Background] Shariat SF, Sfakianos JP, Droller MJ, Karakiewicz PI, Meryn S, Bochner BH. The effect of age and gender on bladder cancer: a critical review of the literature. BJU Int. 2010 Feb;105(3):300-8. doi: 10.1111/j.1464-410X.2009.09076.x. Epub 2009 Nov 13. PMID 19912200
- [Background] Salinas-Sanchez AS, Lorenzo-Romero JG, Gimenez-Bachs JM, Sanchez-Sanchez F, Donate-Moreno MJ, Rubio-Del-Campo A, Hernandez-Millan IR, Segura-Martin M, Atienzar-Tobarra M, Escribano-Martinez J. Implications of p53 gene mutations on patient survival in transitional cell carcinoma of the bladder: a long-term study. Urol Oncol. 2008 Nov-Dec;26(6):620-6. doi: 10.1016/j.urolonc.2007.07.011. Epub 2008 Mar 4. PMID 18367096
- [Background] George B, Datar RH, Wu L, Cai J, Patten N, Beil SJ, Groshen S, Stein J, Skinner D, Jones PA, Cote RJ. p53 gene and protein status: the role of p53 alterations in predicting outcome in patients with bladder cancer. J Clin Oncol. 2007 Dec 1;25(34):5352-8. doi: 10.1200/JCO.2006.10.4125. PMID 18048815
- [Background] Kim PH, Cha EK, Sfakianos JP, Iyer G, Zabor EC, Scott SN, Ostrovnaya I, Ramirez R, Sun A, Shah R, Yee AM, Reuter VE, Bajorin DF, Rosenberg JE, Schultz N, Berger MF, Al-Ahmadie HA, Solit DB, Bochner BH. Genomic predictors of survival in patients with high-grade urothelial carcinoma of the bladder. Eur Urol. 2015 Feb;67(2):198-201. doi: 10.1016/j.eururo.2014.06.050. Epub 2014 Aug 1. PMID 25092538
- [Background] Aljabery F, Shabo I, Gimm O, Jahnson S, Olsson H. The expression profile of p14, p53 and p21 in tumour cells is associated with disease-specific survival and the outcome of postoperative chemotherapy treatment in muscle-invasive bladder cancer. Urol Oncol. 2018 Dec;36(12):530.e7-530.e18. doi: 10.1016/j.urolonc.2018.05.025. Epub 2018 Oct 24. PMID 30539751
- [Background] Wu G, Wang F, Li K, Li S, Zhao C, Fan C, Wang J. Significance of TP53 mutation in bladder cancer disease progression and drug selection. PeerJ. 2019 Dec 16;7:e8261. doi: 10.7717/peerj.8261. eCollection 2019. PMID 31871844
- [Background] Stadler WM, Lerner SP, Groshen S, Stein JP, Shi SR, Raghavan D, Esrig D, Steinberg G, Wood D, Klotz L, Hall C, Skinner DG, Cote RJ. Phase III study of molecularly targeted adjuvant therapy in locally advanced urothelial cancer of the bladder based on p53 status. J Clin Oncol. 2011 Sep 1;29(25):3443-9. doi: 10.1200/JCO.2010.34.4028. Epub 2011 Aug 1. PMID 21810677
- [Background] Knowles MA, Hurst CD. Molecular biology of bladder cancer: new insights into pathogenesis and clinical diversity. Nat Rev Cancer. 2015 Jan;15(1):25-41. doi: 10.1038/nrc3817. PMID 25533674
- [Background] Yang Z, Zhang R, Ge Y, Qin X, Kang X, Wang Y, Zhang X, Song C, Quan X, Wang H, Chen H, Li C. Somatic FGFR3 Mutations Distinguish a Subgroup of Muscle-Invasive Bladder Cancers with Response to Neoadjuvant Chemotherapy. EBioMedicine. 2018 Sep;35:198-203. doi: 10.1016/j.ebiom.2018.06.011. Epub 2018 Jun 22. PMID 29941343
- [Background] Solomon DA, Kim JS, Bondaruk J, Shariat SF, Wang ZF, Elkahloun AG, Ozawa T, Gerard J, Zhuang D, Zhang S, Navai N, Siefker-Radtke A, Phillips JJ, Robinson BD, Rubin MA, Volkmer B, Hautmann R, Kufer R, Hogendoorn PC, Netto G, Theodorescu D, James CD, Czerniak B, Miettinen M, Waldman T. Frequent truncating mutations of STAG2 in bladder cancer. Nat Genet. 2013 Dec;45(12):1428-30. doi: 10.1038/ng.2800. Epub 2013 Oct 13. PMID 24121789
- [Background] Zhu G, Pei L, Li Y, Gou X. EP300 mutation is associated with tumor mutation burden and promotes antitumor immunity in bladder cancer patients. Aging (Albany NY). 2020 Feb 3;12(3):2132-2141. doi: 10.18632/aging.102728. Epub 2020 Feb 3. PMID 32012118
- [Background] Cao Q, Wang C, Ding Y, Xu D, Qian S, Shen H, Qi J. ARID1A upregulation predicts better survival in patients with urothelial bladder carcinoma. J Int Med Res. 2020 Apr;48(4):300060519895687. doi: 10.1177/0300060519895687. Epub 2019 Dec 31. PMID 31891283
- [Background] Wezel F, Vallo S, Roghmann F; Young Academic Urologist Urothelial Carcinoma Group of the European Association of Urology. Do we have biomarkers to predict response to neoadjuvant and adjuvant chemotherapy and immunotherapy in bladder cancer? Transl Androl Urol. 2017 Dec;6(6):1067-1080. doi: 10.21037/tau.2017.09.18. PMID 29354494
- [Background] Kuang S, Li H, Feng J, Xu S, Le Y. Correlation of BRCA2 gene mutation and prognosis as well as variant genes in invasive urothelial carcinoma of the bladder. Cancer Biomark. 2019;25(2):203-212. doi: 10.3233/CBM-182379. PMID 31045513
- [Background] Nickerson ML, Dancik GM, Im KM, Edwards MG, Turan S, Brown J, Ruiz-Rodriguez C, Owens C, Costello JC, Guo G, Tsang SX, Li Y, Zhou Q, Cai Z, Moore LE, Lucia MS, Dean M, Theodorescu D. Concurrent alterations in TERT, KDM6A, and the BRCA pathway in bladder cancer. Clin Cancer Res. 2014 Sep 15;20(18):4935-48. doi: 10.1158/1078-0432.CCR-14-0330. PMID 25225064
- [Background] Plimack ER, Dunbrack RL, Brennan TA, Andrake MD, Zhou Y, Serebriiskii IG, Slifker M, Alpaugh K, Dulaimi E, Palma N, Hoffman-Censits J, Bilusic M, Wong YN, Kutikov A, Viterbo R, Greenberg RE, Chen DY, Lallas CD, Trabulsi EJ, Yelensky R, McConkey DJ, Miller VA, Golemis EA, Ross EA. Defects in DNA Repair Genes Predict Response to Neoadjuvant Cisplatin-based Chemotherapy in Muscle-invasive Bladder Cancer. Eur Urol. 2015 Dec;68(6):959-67. doi: 10.1016/j.eururo.2015.07.009. Epub 2015 Aug 1. PMID 26238431
- [Background] Yin M, Grivas P, Wang QE, Mortazavi A, Emamekhoo H, Holder SL, Drabick JJ, Woo MS, Pal S, Vasekar M, Folefac E, Clinton SK, Monk P, Joshi M. Prognostic Value of DNA Damage Response Genomic Alterations in Relapsed/Advanced Urothelial Cancer. Oncologist. 2020 Aug;25(8):680-688. doi: 10.1634/theoncologist.2019-0851. Epub 2020 May 13. PMID 32275806
- [Background] Fraune C, Simon R, Hube-Magg C, Makrypidi-Fraune G, Kahler C, Kluth M, Hoflmayer D, Buscheck F, Dum D, Luebke AM, Burandt E, Clauditz TS, Wilczak W, Sauter G, Steurer S. MMR deficiency in urothelial carcinoma of the bladder presents with temporal and spatial homogeneity throughout the tumor mass. Urol Oncol. 2020 May;38(5):488-495. doi: 10.1016/j.urolonc.2019.12.012. Epub 2020 Feb 14. PMID 32067846
- [Background] Baras AS, Drake C, Liu JJ, Gandhi N, Kates M, Hoque MO, Meeker A, Hahn N, Taube JM, Schoenberg MP, Netto G, Bivalacqua TJ. The ratio of CD8 to Treg tumor-infiltrating lymphocytes is associated with response to cisplatin-based neoadjuvant chemotherapy in patients with muscle invasive urothelial carcinoma of the bladder. Oncoimmunology. 2016 Feb 18;5(5):e1134412. doi: 10.1080/2162402X.2015.1134412. eCollection 2016 May. PMID 27467953
- [Background] Bellmunt J, Mullane SA, Werner L, Fay AP, Callea M, Leow JJ, Taplin ME, Choueiri TK, Hodi FS, Freeman GJ, Signoretti S. Association of PD-L1 expression on tumor-infiltrating mononuclear cells and overall survival in patients with urothelial carcinoma. Ann Oncol. 2015 Apr;26(4):812-817. doi: 10.1093/annonc/mdv009. Epub 2015 Jan 18. PMID 25600565
- [Background] Li H, Zhang Q, Shuman L, Kaag M, Raman JD, Merrill S, DeGraff DJ, Warrick JI, Chen G. Evaluation of PD-L1 and other immune markers in bladder urothelial carcinoma stratified by histologic variants and molecular subtypes. Sci Rep. 2020 Jan 29;10(1):1439. doi: 10.1038/s41598-020-58351-6. PMID 31996725
- [Background] Topalian SL, Taube JM, Anders RA, Pardoll DM. Mechanism-driven biomarkers to guide immune checkpoint blockade in cancer therapy. Nat Rev Cancer. 2016 May;16(5):275-87. doi: 10.1038/nrc.2016.36. Epub 2016 Apr 15. PMID 27079802
- [Background] Huang HS, Su HY, Li PH, Chiang PH, Huang CH, Chen CH, Hsieh MC. Prognostic impact of tumor infiltrating lymphocytes on patients with metastatic urothelial carcinoma receiving platinum based chemotherapy. Sci Rep. 2018 May 10;8(1):7485. doi: 10.1038/s41598-018-25944-1. PMID 29748589
- [Background] Yu A, Mansure JJ, Solanki S, Siemens DR, Koti M, Dias ABT, Burnier MM, Brimo F, Kassouf W. Presence of lymphocytic infiltrate cytotoxic T lymphocyte CD3+, CD8+, and immunoscore as prognostic marker in patients after radical cystectomy. PLoS One. 2018 Oct 11;13(10):e0205746. doi: 10.1371/journal.pone.0205746. eCollection 2018. PMID 30308033
- [Background] Zhang S, Wang J, Zhang X, Zhou F. Tumor-infiltrating CD8+ lymphocytes predict different clinical outcomes in organ- and non-organ-confined urothelial carcinoma of the bladder following radical cystectomy. PeerJ. 2017 Oct 13;5:e3921. doi: 10.7717/peerj.3921. eCollection 2017. PMID 29043112
- [Background] Kim HS, Ku JH. Prognostic impact of tumor infiltrating lymphocytes in bladder urothelial carcinoma. Transl Androl Urol. 2019 Jul;8(Suppl 3):S291-S292. doi: 10.21037/tau.2019.04.02. No abstract available. PMID 31392149
- [Background] Liu H, Ye T, Yang X, Lv P, Wu X, Zhou H, Lu H, Tang K, Ye Z. Predictive and Prognostic Role of PD-L1 in Urothelial Carcinoma Patients with Anti-PD-1/PD-L1 Therapy: A Systematic Review and Meta-Analysis. Dis Markers. 2020 Jun 27;2020:8375348. doi: 10.1155/2020/8375348. eCollection 2020. PMID 32685057